CLINICAL TRIAL: NCT03900832
Title: Effects of Heating on Exercise Pressor Reflex in Peripheral Artery Disease: Exercise Ability
Acronym: EPR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jian Cui, Associate Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00005798
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: PAD
Keywords: exercise; blood pressure response; heating
MeSH Terms: conditions — Motor Activity | interventions — Heating

STUDY DESIGN:
Intervention Model Description: The investigators will examine (using a prospective observational design) if heating will affect walking ability, blood pressure and heart rate responses in PAD patients. Each subject will serve as their own control. Additionally, we will compare these responses between PAD patients and healthy controls subjects.
Who Masked: Outcomes Assessor
Masking Description: Subjects will be aware if they are being heated or not, but data analysis process is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- PAD without heating (Placebo Comparator): Subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Without Heating; Other: Gardner walking protocol
- PAD warm bath (Experimental): Subjects will take a warm bath. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Warm Bath; Other: Gardner walking protocol
- PAD neutral bath (Placebo Comparator): Subjects will take a neutral bath. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Neutral Bath; Other: Gardner walking protocol
- PAD heating suit (Experimental): Whole body heating with the suit will be performed. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Heating Suit; Other: Gardner walking protocol
- PAD lower limb warm water immersion (Experimental): Subjects will place their lower legs in warm water. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Lower limb warm water immersion; Other: Gardner walking protocol
- Healthy subjects without heating (Placebo Comparator): Subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Without Heating; Other: Gardner walking protocol
- Healthy subjects warm bath (Experimental): Subjects will take a warm bath. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Warm Bath; Other: Gardner walking protocol
- Healthy subjects neutral bath (Placebo Comparator): Subjects will take a neutral bath. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Neutral Bath; Other: Gardner walking protocol
- Healthy subjects heat suit (Experimental): Whole body heating with the suit will be performed. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Heating Suit; Other: Gardner walking protocol
- Healthy subjects lower limb immersion (Experimental): Subjects will place their lower legs in warm water. Then, subjects will walk on a treadmill using the Gardner protocol until the patient says they want to stop. BP, HR and NIRS will be continuously measured during Gardner protocol. Skin blood flow, skin temperature and BP will be measured in the supine position before and after the Gardner protocol.
  Interventions: Other: Lower limb warm water immersion; Other: Gardner walking protocol

INTERVENTIONS:
Other: Without Heating — Subject will complete walking protocol without any heating procedure
  Arms: Healthy subjects without heating; PAD without heating
Other: Warm Bath — Subjects will sit in a warm bathtub with water up to their shoulders, while one arm will be out of water for BP and HR measurement. The water temperature and internal temperature (Tcore), BP and HR will be measured throughout the bath.
  The water temperature will be controlled between 38-41°C. Subjects will remain in the tub for ≤ 30 minutes. If the HR increases more than 15 -20 bpm, or a significant BP drop occurs (e.g. BP >20 mmHg), the subject will be removed from the bath even if the time is <30 min.
  Arms: Healthy subjects warm bath; PAD warm bath
Other: Neutral Bath — Subjects will sit in a warm bathtub with water up to their shoulders, while one arm will be out of water for BP and HR measurement. The water temperature and internal temperature (Tcore), BP and HR will be measured throughout the bath.
  The water temperature will be controlled between 35 - 37°C. Subjects will remain in the tub for ≤ 30 minutes.
  Arms: Healthy subjects neutral bath; PAD neutral bath
Other: Heating Suit — The mean skin temperature Tsk will be controlled with a water-perfused suit worn by subjects. Whole-body heating will be accomplished by perfusing warm water (~ 45 - 50 °C) through the suit to elevate the Tsk to ≤ 38 °C (100 oF). Warm water is through plastic tubes, and subjects' skin will not directly touch warm water. The heating will be continued until the ∆Tcore reaches ~ 0. 6 - 1.0 °C. This may take approximately 60 - 90 min.
  Arms: Healthy subjects heat suit; PAD heating suit
Other: Lower limb warm water immersion — Subjects will sit on a chair and put their lower legs and feet in a bucket with warm water. The water level will be just below the knees (depth of approximately 40 cm). The water temperature will be monitored and controlled at ~38 - 42 °C throughout the 30 minutes. BP, HR, Tcore, the skin temperature and skin blood flow (e.g. on a thigh and/or forearm) will be measured before, during and after the lower limbs warm water immersion.
  Arms: Healthy subjects lower limb immersion; PAD lower limb warm water immersion
Other: Gardner walking protocol — The Gardner protocol begins at 2 mph and 0% grade for 2 minutes. The grade increases by 2% every 2 minutes (the speed remains 2 mph) until the subject says they want to stop or 22 minutes maximum. BP and HR will also be measured throughout the protocol.

SUMMARY:
The study objectives of this projects are to examine the hypothesis that the sympathetic and blood pressure responses to exercise will be attenuated during and after heat exposure in patients with peripheral artery disease, via altering the sensitivity of the muscle afferent receptors.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects 8-12 million Americans and its cardinal symptom is leg pain during exercise, termed "intermittent claudication". The diagnosis of PAD involves measuring the ankle-brachial index (ABI, i.e. the systolic pressure in the ankle divided by the systolic pressure in the arm); values below 0.9 are indicative of large vessel obstruction. Intermittent claudication is the most common symptom of this disease and it regularly occurs during exercise/physical activity but is relieved promptly by rest. Previous studies suggest that as the exercise pressor reflex is activated in patients with PAD, BP and heart rate (HR) are exaggerated. The BP rises during walking in the PAD patients were significantly greater than that seen in healthy control subjects. A recent human study from our group further indicates that an early BP response occurred during plantar flexion exercise before claudication was noted by the subjects, which may suggest that the accentuated BP response was due to an augmented muscle mechanoreflex in PAD. Moreover, another recent study from our group also showed that PAD patients have augmented renal vasoconstriction during plantar flexion exercise.

It has been shown that exercise has benefits for patients with PAD. However, exercise becomes limited due to the pain and fatigue associated with the disease. Moreover, the augmented pressor response to exercise in PAD may increase the risk for the end organ damage (e.g. brain and/or heart). Thus, finding alternate/complimentary interventions that modulate the cardiovascular system and autonomic nervous system, and can be tolerated by the patients, would be beneficial.

One possible intervention is heat exposure, since acute bouts of exercise and acute heat exposure have similar acute effects on both the autonomic and cardiovascular systems. For example, both exercise and heat exposure increase body temperature, increase HR, increase cardiac output (CO), increase left ventricular ejection fraction (EF), and enhance myocardial function. In the peripheral circulation, both exercise and heat exposure increase limb blood flow , muscle blood flow, and skin blood flow. Moreover, recent studies suggest that whole body exposure improves the endothelium function in PAD patients (e.g. activates endothelial progenitor cells CD34+).

However, the effect of heat treatment on the ability of walking of PAD patients has not been examined. Moreover, it is unknown if heating can normalize/decrease the accentuated the pressor responses to exercise in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Capable of giving informed consent
* Any race or ethnicity
* Men and women age 21- 85 years (inclusive)
* Fluent in written and spoken English

Patients with peripheral arterial disease (PAD)

* Diagnosed with PAD (i.e., ankle-brachial index below 0.9)
* Fontaine stage II or less - no pain while resting
* Satisfactory history and physical exam

Healthy subjects

* Satisfactory history and physical examination
* Free of acute medical conditions

Exclusion Criteria:

For patients with PAD and Healthy subjects

* Age < 21 years
* Pregnant or nursing women
* Decisional impairment
* Prisoners

For patients with PAD

* History of CAD with symptoms of unstable angina or myocardial infarction (<6 months)
* History of epilepsy or seizure disorders

For healthy subjects

• Any other chronic diseases (heart, lung, neuromuscular disease or diabetes)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Walking time in minutes | Recording walking time to fatigue (up to 22 minutes maximum) during of every 3-4 hour study visit.
  Walking time on treadmill using Gardner protocol
Blood pressure in mmHg | Recorded continuously during the 3-4 hour study visit
  Cuffs placed on a finger and arm will monitor blood pressure.
Heart Rate in beats per minute | Recorded continuously during the 3-4 hour study visit
  Electrocardiogram (ECG) patches attached to a Cardiocap will monitor heart rat

SECONDARY OUTCOMES:
Internal Temperature in degrees C | Recorded continuously during the 3-4 hour study visit
  The internal temperature (Tcore) will be measured from the stomach/intestines via a telemetry pill swallowed by subjects.
Near infrared spectroscopy (NIRS) in arbitrary units | Recorded continuously during the 3-4 hour study visit
  This system is designed specifically for non-invasive measurements of muscle tissue. The system measures the tissue saturation of the investigated muscle, called the 'tissue saturation index' (TSI).

CONTACTS AND LOCATIONS:
Overall Officials: Jian Cui, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui J, Blaha C, Sinoway LI. Whole body heat stress attenuates the pressure response to muscle metaboreceptor stimulation in humans. J Appl Physiol (1985). 2016 Nov 1;121(5):1178-1186. doi: 10.1152/japplphysiol.00212.2016. Epub 2016 Oct 7. PMID 27763873
- [Background] Cui J, Blaha C, Moradkhan R, Gray KS, Sinoway LI. Muscle sympathetic nerve activity responses to dynamic passive muscle stretch in humans. J Physiol. 2006 Oct 15;576(Pt 2):625-34. doi: 10.1113/jphysiol.2006.116640. Epub 2006 Jul 27. PMID 16873399
- [Background] Cui J, Boehmer J, Blaha C, Sinoway LI. Muscle sympathetic nerve activity response to heat stress is attenuated in chronic heart failure patients. Am J Physiol Regul Integr Comp Physiol. 2017 Jun 1;312(6):R873-R882. doi: 10.1152/ajpregu.00355.2016. Epub 2017 Mar 22. PMID 28330967
- [Background] Cui J, Muller MD, Blaha C, Kunselman AR, Sinoway LI. Seasonal variation in muscle sympathetic nerve activity. Physiol Rep. 2015 Aug;3(8):e12492. doi: 10.14814/phy2.12492. PMID 26265752